CLINICAL TRIAL: NCT06046625
Title: The Needs and Preferences of Patients With High-risk Cutaneous Squamous Cell Carcinomas in the Head Neck Region: a Qualitative Approach
Brief Title: Needs and Preferences of Patients With Head-neck Cutaneous SCC
Status: Active, not recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 2021-2765
Record Dates: First submitted 2023-08-18; First posted 2023-09-21 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Cutaneous Squamous Cell Carcinoma of the Head and Neck; Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck; Squamous Cell Carcinoma of the Head and Neck; Skin Cancer; Patient Satisfaction; High-Risk Cancer; Preference, Patient; Decision Making; Interview
Keywords: Patient experience; Patients need; Semi-structured; Professionals; Experience; Needs
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Skin Neoplasms; Patient Satisfaction; Patient Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Head-neck cutaneous Squamous cell carcinomas: Patients with high risk cutaneous squamous cell carcinoma in the head neck region, receiving regular multidisciplinary care.
  Interventions: Other: Regular care with additional administration of a semi-structured interview

INTERVENTIONS:
Other: Regular care with additional administration of a semi-structured interview — Patients receiving regular care. In addition, a semi-structured interview is conducted.
  The semi-structured interviews take place once after completion of the care pathway (after all appointments for check-ups associated with the treatment). The interview contains questions about the experience of patients with the care, the needs in this care, the experiences with the information received, the support/guidance, the turnaround time, the treatment received and areas for improvement.

SUMMARY:
The care of patients with high-risk cutaneous squamous cell carcinomas in the head-neck area is complex and requires a multidisciplinary approach. A key component in this care is the need and experience of patients. However, studies on the experiences and needs of patients with high-risk cutaneous squamous cell carcinomas in the head-neck region are lacking.

DETAILED DESCRIPTION:
Cutaneous squamous cell carcinoma (cSCC) is the second most common form of skin cancer worldwide after basal cell carcinoma. It involves approximately 20% of all cutaneous malignancies and its incidence is still increasing. In 2020, nearly 15,000 cSCCs were reported in the Netherlands, of which approximately 50% concerned patients aged 75 years or older. UV radiation is the main risk factor for development of a cSCC, therefore the majority of cSCCs are localized to the sun-exposed skin in the head-neck region. cSCCs have a metastatic rate of 2.6-5% and recurrence rate of 1.9-3.7%, with rates increasing in high-risk cSCCs. The increasing incidence, advanced age, the (often) high-risk localization in the head-neck area (given functional and cosmetic importance) and the possible high risk of metastasis result in complex care, especially in stage T2 to T4 cSCCs, also known as high-risk cSCCs.

In this complex care, care pathways offer an excellent opportunity to improve multidisciplinary communication, patient satisfaction, quality and efficiency of care. In this, the experiences and needs of patients are of great importance. Previous research on the experiences and needs of patients with skin cancer is limited and particularly focused on melanomas. In 2017, a qualitative systematic review of the experiences and needs of patients with skin cancer found only two studies examining cSCCs. These studies showed that patients perceived clear information, attention to psychosocial aspects and attention to prevention as important.

In 2019, a study of the needs and experiences of patients with keratinocyte carcinomas, conducted through focus groups, showed similar results. Non of these studies examined cSCCs exclusively, nor did they differentiate by location. However, this appears to be relevant, because of the higher impact on the quality of life of patients with skin cancer in visible locations.

Additionally, studies have been conducted into shared-decision making as part of multidisciplinary care. Complex cases are currently often discussed multidisciplinary. However, several studies describe that such a multidisciplinary approach can impede multidisciplinary decision-making because the patient's perspective is often missing. Studies on the experience of patients with cSCCs in the head neck region are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a cSCC, located in the head-neck region
* who visited the multidisciplinary head-neck team of the Maastricht University Medical Center+
* who already received treatment for their cSCC
* who gave informed consent for participation

Exclusion Criteria:

- patients who are cognitively impaired for participation in an interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, over 18 years of age, clinically diagnosed with a cutaneous squamous cell carcinoma localized in the head and neck area, seen in the MUMC+ at the multidisciplinary head-neck consultation of the department of dermatology, who have already been treated for this cSCC and are willing to participate in the study will be included. If the patient is cognitively unable to participate in the interview, alternatively, a representative may participate in the interview.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Themes patients | Through study completion, an average of 1 year
  The emerging themes of patient needs an experiences in the care of cutaneous squamous cell carcinoma in the head-neck region.
Themes professionals | Through study completion, an average of 1 year
  The emerging themes of professionals' needs in the care of patients with cutaneous squamous cell carcinoma in the head-neck area.

SECONDARY OUTCOMES:
Association themes and patient/tumor characteristics | Through study completion, an average of 1 year
  The associations between the emerging themes and baseline characteristics (such as gender, age, marital status, education level, world health organisation performance status, informal care, history of skin cancer, co-occurrence of other skin cancers) and tumor characteristics (such as stage of cSCC, differentiation, type of treatment).
Association themes and professional characteristics | Through study completion, an average of 1 year
  The associations between the emerging themes and characteristics of professionals (gender, age, type of specialty, number of years working as a specialist, number of years of experience within head and neck working group).

CONTACTS AND LOCATIONS:
Overall Officials: K Mosterd, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center+, Maastricht, Netherlands

REFERENCES:
- [Background] Fania L, Didona D, Di Pietro FR, Verkhovskaia S, Morese R, Paolino G, Donati M, Ricci F, Coco V, Ricci F, Candi E, Abeni D, Dellambra E. Cutaneous Squamous Cell Carcinoma: From Pathophysiology to Novel Therapeutic Approaches. Biomedicines. 2021 Feb 9;9(2):171. doi: 10.3390/biomedicines9020171. PMID 33572373
- [Background] Stratigos AJ, Garbe C, Dessinioti C, Lebbe C, Bataille V, Bastholt L, Dreno B, Fargnoli MC, Forsea AM, Frenard C, Harwood CAlpha, Hauschild A, Hoeller C, Kandolf-Sekulovic L, Kaufmann R, Kelleners-Smeets NW, Malvehy J, Del Marmol V, Middleton MR, Moreno-Ramirez D, Pellecani G, Peris K, Saiag P, van den Beuken-van Everdingen MHJ, Vieira R, Zalaudek I, Eggermont AMM, Grob JJ; European Dermatology Forum (EDF), the European Association of Dermato-Oncology (EADO) and the European Organization for Research and Treatment of Cancer (EORTC). European interdisciplinary guideline on invasive squamous cell carcinoma of the skin: Part 1. epidemiology, diagnostics and prevention. Eur J Cancer. 2020 Mar;128:60-82. doi: 10.1016/j.ejca.2020.01.007. Epub 2020 Feb 26. PMID 32113941
- [Background] Stern RS; PUVA Follow-Up Study. The risk of squamous cell and basal cell cancer associated with psoralen and ultraviolet A therapy: a 30-year prospective study. J Am Acad Dermatol. 2012 Apr;66(4):553-62. doi: 10.1016/j.jaad.2011.04.004. Epub 2012 Jan 20. PMID 22264671
- [Background] Kallini JR, Hamed N, Khachemoune A. Squamous cell carcinoma of the skin: epidemiology, classification, management, and novel trends. Int J Dermatol. 2015 Feb;54(2):130-40. doi: 10.1111/ijd.12553. Epub 2014 Nov 27. PMID 25428226
- [Background] Klaus Wolff RAJ, Arturo P. Saavedra, Ellen K. Roh. SECTION 11: PRECANCEROUS LESIONS AND CUTANEOUS CARCINOMAS. Fitzpatrick's Color Atlas and Synopsis of Clinical Dermatology. Eigth edition ed: McGraw-Hill Education; 2017
- [Background] Que SKT, Zwald FO, Schmults CD. Cutaneous squamous cell carcinoma: Incidence, risk factors, diagnosis, and staging. J Am Acad Dermatol. 2018 Feb;78(2):237-247. doi: 10.1016/j.jaad.2017.08.059. PMID 29332704
- [Background] Mourouzis C, Boynton A, Grant J, Umar T, Wilson A, Macpheson D, Pratt C. Cutaneous head and neck SCCs and risk of nodal metastasis - UK experience. J Craniomaxillofac Surg. 2009 Dec;37(8):443-7. doi: 10.1016/j.jcms.2009.07.007. Epub 2009 Aug 27. PMID 19713116
- [Background] Brantsch KD, Meisner C, Schonfisch B, Trilling B, Wehner-Caroli J, Rocken M, Breuninger H. Analysis of risk factors determining prognosis of cutaneous squamous-cell carcinoma: a prospective study. Lancet Oncol. 2008 Aug;9(8):713-20. doi: 10.1016/S1470-2045(08)70178-5. Epub 2008 Jul 9. PMID 18617440
- [Background] Brougham ND, Dennett ER, Cameron R, Tan ST. The incidence of metastasis from cutaneous squamous cell carcinoma and the impact of its risk factors. J Surg Oncol. 2012 Dec;106(7):811-5. doi: 10.1002/jso.23155. Epub 2012 May 16. PMID 22592943
- [Background] Schmults CD, Karia PS, Carter JB, Han J, Qureshi AA. Factors predictive of recurrence and death from cutaneous squamous cell carcinoma: a 10-year, single-institution cohort study. JAMA Dermatol. 2013 May;149(5):541-7. doi: 10.1001/jamadermatol.2013.2139. PMID 23677079
- [Background] Muzic JG, Schmitt AR, Wright AC, Alniemi DT, Zubair AS, Olazagasti Lourido JM, Sosa Seda IM, Weaver AL, Baum CL. Incidence and Trends of Basal Cell Carcinoma and Cutaneous Squamous Cell Carcinoma: A Population-Based Study in Olmsted County, Minnesota, 2000 to 2010. Mayo Clin Proc. 2017 Jun;92(6):890-898. doi: 10.1016/j.mayocp.2017.02.015. Epub 2017 May 15. PMID 28522111
- [Background] van Hoeve JC, Vernooij RWM, Fiander M, Nieboer P, Siesling S, Rotter T. Effects of oncological care pathways in primary and secondary care on patient, professional and health systems outcomes: a systematic review and meta-analysis. Syst Rev. 2020 Oct 25;9(1):246. doi: 10.1186/s13643-020-01498-0. PMID 33100227
- [Background] Bath-Hextall F, Nalubega S, Evans C. The needs and experiences of patients with skin cancer: a qualitative systematic review with metasynthesis. Br J Dermatol. 2017 Sep;177(3):666-687. doi: 10.1111/bjd.15148. Epub 2017 Feb 22. PMID 27775838
- [Background] Winterbottom A, Harcourt D. Patients' experience of the diagnosis and treatment of skin cancer. J Adv Nurs. 2004 Nov;48(3):226-33. doi: 10.1111/j.1365-2648.2004.03191.x. PMID 15488036
- [Background] Bath-Hextall F, Jenkinson C, Kumar A, Leonardi-Bee J, Perkins W, Cox K, Glazebrook C. Longitudinal, mixed method study to look at the experiences and knowledge of non melanoma skin cancer from diagnosis to one year. BMC Dermatol. 2013 Oct 29;13:13. doi: 10.1186/1471-5945-13-13. PMID 24164857
- [Background] van Egmond S, Wakkee M, Droger M, Bastiaens MT, van Rengen A, de Roos KP, Nijsten T, Lugtenberg M. Needs and preferences of patients regarding basal cell carcinoma and cutaneous squamous cell carcinoma care: a qualitative focus group study. Br J Dermatol. 2019 Jan;180(1):122-129. doi: 10.1111/bjd.16900. Epub 2018 Sep 23. PMID 29927480
- [Background] Abedini R, Nasimi M, Noormohammad Pour P, Moghtadaie A, Tohidinik HR. Quality of Life in Patients with Non-melanoma Skin Cancer: Implications for Healthcare Education Services and Supports. J Cancer Educ. 2019 Aug;34(4):755-759. doi: 10.1007/s13187-018-1368-y. PMID 29705894
- [Background] Hamilton DW, Heaven B, Thomson RG, Wilson JA, Exley C. Multidisciplinary team decision-making in cancer and the absent patient: a qualitative study. BMJ Open. 2016 Jul 21;6(7):e012559. doi: 10.1136/bmjopen-2016-012559. PMID 27443554
- [Background] Hahlweg P, Hoffmann J, Harter M, Frosch DL, Elwyn G, Scholl I. In Absentia: An Exploratory Study of How Patients Are Considered in Multidisciplinary Cancer Team Meetings. PLoS One. 2015 Oct 6;10(10):e0139921. doi: 10.1371/journal.pone.0139921. eCollection 2015. PMID 26441328